CLINICAL TRIAL: NCT00551278
Title: GeneSearch™ Breast Lymph Node (BLN) Assay for Molecular Testing Protocol
Brief Title: Validation Study Using the GeneSearch BLN Assay to Test Sentinel Lymph Nodes From Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Janssen Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BLN-US-IU-2006.00
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: sentinel lymph node; metastasis; molecular pathology
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Biological Assay

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of the tissue homogenate and extracted RNA will be retained and may be used for for further testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with previous diagnosis of breast cancer scheduled for sentinel lymph node dissection.
  Interventions: Device: GeneSearch™ Breast Lymph Node (BLN) Assay

INTERVENTIONS:
Device: GeneSearch™ Breast Lymph Node (BLN) Assay — For in vitro diagnostic use only.
  The GeneSearch™ Breast Lymph Node (BLN) Assay is a qualitative, in vitro diagnostic test for the rapid detection of greater than 0.2 mm metastases in nodal tissue removed from sentinel lymph node biopsies of breast cancer patients. Results from the assay can be used to guide the intra-operative or post-operative decision to remove additional lymph nodes.
  Post-operative histological evaluation of permanent sections of the tissue specimen, in accordance with usual diagnostic practice and using the Veridex lymph node cutting scheme, is required.

SUMMARY:
The purpose of this trial is to show adequate assay performance on clinical samples tested in real time at the clinical site.

DETAILED DESCRIPTION:
This study will determine the sensitivity, specificity, negative predictive value, and positive predictive value of the GeneSearch™ BLN Assay in patient samples by comparing its performance to that of the current methods -- permanent section Hematoxylin and Eosin (H&E) staining with IHC. Additional marker testing using probes associated with nodal metastases may be used in the assay performance calculations. The observed performance measures will be compared to those obtained in the larger U.S. registration trial to show that there are no differences in the assay's performance.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of carcinoma of the breast
* Patient scheduled for sentinel lymph node dissection as per standard of care at the clinical site
* 18 years or older
* Female or male, and
* Able and willing to give consent to participate in the study

Exclusion Criteria:

* Patients taking part in other research studies that would interfere with their full participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a previous diagnosis of breast cancer scheduled for sentinel lymph node dissection.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The study will determine the sensitivity, specificity, negative predictive value and positive predictive value of the GeneSearch™ BLN Assay by comparing its performance to permanent section Hematoxylin and Eosin (H&E) staining with IHC. | 1 month

SECONDARY OUTCOMES:
A secondary objective will assess the timing and logistical aspects of introducing a real time molecular test within the pathology lab. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Goulet, MD, Principal Investigator — Indiana University Cancer Pavilion
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States